CLINICAL TRIAL: NCT00601276
Title: Comparative Controlled Clinical Trial of Two Pharmacological Treatments of Pedophilia
Brief Title: Comparison of Two Pharmacological Treatments of Pedophilia
Acronym: PCNET
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); Ministry of Health, France (Other Government); Ministry of Higher Education and Research, France (Other Government)
Responsible Party: Dr Stoleru, Inserm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RBM-0315
Record Dates: First submitted 2007-12-03; First posted 2008-01-28 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2007-12

CONDITIONS: Pedophilia
Keywords: pedophilia; antiandrogens; gonadotropin releasing hormone agonists
MeSH Terms: conditions — Pedophilia | interventions — Leuprolide; Cyproterone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: leuprorelin
- 2 (Active Comparator)
  Interventions: Drug: Cyproterone acetate

INTERVENTIONS:
Drug: leuprorelin — Subcutaneous injection, 3.75 mg every 4 weeks
  Other Names: Enantone
  Arms: 1
Drug: Cyproterone acetate — 2.0 mg/kg/day, tablet, per os
  Other Names: Androcur
  Arms: 2

SUMMARY:
Sexual abuse committed on children is a major public health problem because of its frequency and its severe consequences on the mental health of victims.

Objective: to compare the therapeutic efficacy of cyproterone acetate (CPA) and leuprolide, with the hypothesis that leuprolide will be more effective.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of pedophilia
* high frequency of sexual urges and deviant behavior as demonstrated by a score equal to 8 on the scale of Rösler & Witztum (Rösler & Witztum, 1998) ;
* age: 18-60 years
* informed consent

Exclusion Criteria:

* IQ<70
* schizophrenia, schizoaffective disorder, or delusional disorder
* already receiving one of the tested drugs
* contraindication for one of the tested drugs
* no current or planned incarceration

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Questionnaire on sexual behavior | prospective

SECONDARY OUTCOMES:
Recidivism | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Serge Stoleru, MD, PHD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (4):
- France (4):
  - Federation d'Endocrinologie, Hopital NeuroCardiologique, Bron
  - Centre MédicoPsychologique CMPG21, EPS Perray Vaucluse, Paris
  - Service de Psychiatrie, Hopital Foch, Suresnes
  - SMPR, Hopital Paul Guiraud, Villejuif

REFERENCES:
- [Derived] Moulier V, Fonteille V, Pelegrini-Issac M, Cordier B, Baron-Laforet S, Boriasse E, Durand E, Stoleru S. A pilot study of the effects of gonadotropin-releasing hormone agonist therapy on brain activation pattern in a man with pedophilia. Int J Offender Ther Comp Criminol. 2012 Feb;56(1):50-60. doi: 10.1177/0306624X10392191. Epub 2011 Apr 24. PMID 21518701